CLINICAL TRIAL: NCT04049799
Title: Medically-supervised Withdrawal vs. Agonist Maintenance in the Treatment of Pregnant Women With Opioid Use Disorder: Maternal, Fetal, and Neonatal Outcomes
Brief Title: Maternal Opioid Treatment: Human Experimental Research - Data Yield Appropriate Decisions
Acronym: MOTHER DYAD
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Virginia Commonwealth University (Other); Mountain Area Health Education Center (Unknown); Johns Hopkins University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sarah Heil, Professor, University of Vermont
Other Study IDs: STUDY00000166; R01DA047867 (NIH)
Record Dates: First submitted 2019-07-23; First posted 2019-08-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Opioid-use Disorder; Opioid Withdrawal; Neonatal Abstinence Syndrome; Neonatal Opioid Withdrawal Syndrome
MeSH Terms: conditions — Opioid-Related Disorders; Neonatal Abstinence Syndrome | interventions — Inactivation, Metabolic; Maintenance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medically-supervised withdrawal (MSW)
  Interventions: Other: Medically-supervised withdrawal; Behavioral: Comprehensive clinical care
- Opioid agonist treatment (OAT)
  Interventions: Other: Opioid agonist treatment; Behavioral: Comprehensive clinical care

INTERVENTIONS:
Other: Medically-supervised withdrawal — 6-8 day withdrawal with buprenorphine/naloxone
  Other Names: Detoxification
  Groups: Medically-supervised withdrawal (MSW)
Other: Opioid agonist treatment — Induction and maintenance with buprenorphine/naloxone
  Other Names: Maintenance
  Groups: Opioid agonist treatment (OAT)
Behavioral: Comprehensive clinical care — Obstetrical visits, counseling, case management, psychiatry services, and urine drug screening

SUMMARY:
This study will compare medically-supervised withdrawal (MSW, 'detoxification') to opioid agonist treatment (OAT, 'maintenance') with buprenorphine for pregnant women with opioid use disorder in terms of maternal, fetal, and neonatal outcomes. Outcomes will be assessed during pregnancy, at birth and for 12 months postpartum. This study has the potential to impact health service policy and practices in terms of the treatment options of pregnant women with opioid use disorder.

DETAILED DESCRIPTION:
Some inclusion/exclusion criteria are purposely omitted at this time to preserve scientific integrity. They will be included after the trial is complete.

ELIGIBILITY:
Inclusion Criteria:

* Be ages 18 to 41, inclusive
* Have a single fetus pregnancy between 6-30 weeks estimated gestational age
* Willing to participate in the study

Exclusion Criteria:

* Non-English speaking

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women seeking treatment for opioid use disorder
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Proportion of mothers who discontinued 1st treatment choice prior to delivery | Antepartum period
Proportion of mothers engaged in treatment at delivery | Antepartum period
  Behavior health treatment or medical treatment in past 21 days
Proportion of mothers with illicit substance use at delivery | At delivery
  Positive vs. negative for any illicit substance in the urine
Proportion of mother-child dyads with delivery complications | At delivery
  Yes vs. no code for the presence or absence of delivery complications such as uterine rupture, placental abruption, low birth weight, chorioamnionitis, and meconium staining
Proportion of neonates receiving medication treatment for neonatal abstinence syndrome (NAS) | At hospital discharge, an average of 10 days after delivery
  Yes vs. no
Total average amount of medication given to treat NAS | At hospital discharge, an average of 10 days after delivery
  Morphine Equivalent Dose in mg
Total average length of neonatal hospital stay | At hospital discharge, an average of 10 days after delivery
  Days

CONTACTS AND LOCATIONS:
Overall Officials: Sarah H Heil, PhD, Principal Investigator — University of Vermont
Locations (4):
- United States (4):
  - Mountain Area Health Education Center, Asheville, North Carolina
  - UNC Chapel Hill Horizons, Chapel Hill, North Carolina
  - University of Vermont, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia